CLINICAL TRIAL: NCT00553644
Title: A Phase II Trial of Bortezomib (NSC #681239) + Lenalidomide (Revlimid™, CC-5013) (NSC #703813) for Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Bortezomib and Lenalidomide in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00483; NCI-2009-00483 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000573827; CALGB 50501 (Other: Alliance for Clinical Trials in Oncology); CALGB-50501 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; Lenalidomide

ARMS (1):
- Treatment (bortezomib, lenalidomide) (Experimental): Patients receive induction therapy comprising bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and lenalidomide PO QD on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response as best response after completion of induction therapy receive maintenance therapy comprising bortezomib IV on days 1 and 8 and lenalidomide PO QD on days 1-14. Treatment repeats every 21 days for up to 6 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies how well bortezomib and lenalidomide work in treating patients with mantle cell lymphoma that has come back after a period of improvement (refractory) or is not responding to treatment (refractory). Bortezomib may also stop the growth of cancer cells by blocking some proteins needed for cell growth. Lenalidomide may stimulate the immune system to kill cancer cells and may also block the growth of new blood vessels necessary for cell growth. Giving bortezomib with lenalidomide may be an effective treatment for relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response (complete response [CR] and partial response [PR]) rate and the complete response (CR) rate to bortezomib + lenalidomide therapy in patients with relapsed or refractory mantle cell lymphoma.

SECONDARY OBJECTIVES:

I. To determine the time to progression after therapy with bortezomib + lenalidomide in patients with relapsed or refractory mantle cell lymphoma.

II. To determine the disease-free survival and overall survival after therapy with bortezomib + lenalidomide in patients with relapsed or refractory mantle cell lymphoma.

OUTLINE:

Patients receive induction therapy comprising bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11 and lenalidomide orally (PO) once daily (QD) on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response as best response after completion of induction therapy receive maintenance therapy comprising bortezomib IV on days 1 and 8 and lenalidomide PO QD on days 1-14. Treatment repeats every 21 days for up to 6 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented mantle cell lymphoma, with the following immunophenotypic characteristics: cluster of differentiation (CD)5+, CD23-, cyclin D1+; this may be from an initial diagnostic biopsy, or one obtained at time of relapse

  * Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies; fine needle aspirates are not acceptable
  * Failure to submit pathology specimens within 60 days of patient registration will be considered a major protocol violation
* Institutional flow cytometry or immunohistochemistry must confirm CD5 antigen expression, lack of CD23 antigen expression, and expression of cyclin D1
* Prior therapy with at least one regimen, which may have been single agent or multi-agent, and consisted of traditional cytotoxic agents and/or biologic agents; patient may not have received prior bortezomib or lenalidomide therapy; patient must have progressive disease or refractory disease following that initial regimen(s); refractory disease will be defined as stable disease (SD) or progressive disease (PD) as best response to prior therapy, or CR or PR as initial response followed by disease progression within 6 months
* Prior autologous, but not allogeneic, stem cell transplant is allowed
* No corticosteroids within two weeks prior to study, except for maintenance therapy for a non-malignant disease; maintenance therapy dose may not exceed 20 mg/day prednisone or equivalent
* No prior radioimmunotherapy within 12 months of study entry
* No >= grade 3 peripheral neuropathy within a month prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm by physical exam, computed tomography (CT), magnetic resonance imaging (MRI), or conventional radiograph is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions (lesions, if present, should be noted)
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis or pulmonis
  * Bone marrow (involvement by non-Hodgkin lymphoma should be noted)
* No known central nervous system (CNS) involvement by lymphoma
* Patients with human immunodeficiency virus (HIV) infection are eligible, provided they meet the following: CD4+ cell count > 350/mm^3; treatment sensitive HIV and, if on anti-HIV therapy, HIV viral load < 50 copies/mm^3; no history of acquired immunodeficiency syndrome (AIDS)-defining conditions or other HIV-related illnesses; no concurrent zidovudine or stavudine
* Non-pregnant and non-nursing; females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to registration; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure; documentation of counseling is required on Cancer and Leukemia Group B (CALGB) form S-041
* Patients with a recent history (within 3 months of study entry) of deep vein thrombosis (DVT)/pulmonary embolism (PE) are not eligible; patients with a distant history (greater than 3 months before study entry) of DVT/PE are eligible, but must receive either prophylactic aspirin or low molecular weight heparin, unless contraindicated
* Left ventricular ejection fraction (LVEF) >= 45% by multigated acquisition (MUGA) scan or echocardiogram
* No New York Heart Association class III or class IV congestive heart failure at study entry
* No myocardial infarction within the past 6 months of study entry
* No known positivity for hepatitis A, B, or C
* Absolute neutrophil count (ANC) >= 1,000/uL (>= 500/uL if marrow involvement)
* Platelets >= 75,000/uL
* Creatinine =< 1.5 x upper limit of normal (ULN) (unless attributable to non-Hodgkin's lymphoma) and estimated creatinine clearance >= 30 mL/min (patients on dialysis are not eligible)
* Total bilirubin =< 2 x ULN (unless attributable to non-Hodgkin's lymphoma and Gilbert's disease)
* Urine (U)-human chorionic gonadotropin (HCG) or serum HCG negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-11-15 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2014-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Morrison, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (82):
- United States (82):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Hartford Hospital, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - McLeod Regional Medical Center, Florence, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2007 and July 2011, 54 participants were recruited to this study.
Pre-assignment Details: One participant was deemed ineligible and removed for all analyses; therefore, 53 participants were analyzed.
Groups:
- Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy): Patients receive induction therapy comprising bortezomib 1.3mg/m^2 IV over 3-5 seconds on days 1, 4, 8, and 11 and lenalidomide 20 mg/day PO once daily on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response as best response after completion of induction therapy receive maintenance therapy comprising bortezomib 1.3 mg/m^2 IV on days 1 and 8 and lenalidomide 15 mg/day PO once daily on days 1-14. Treatment repeats every 21 days for up to 6 years in the absence of disease progression or unacceptable toxicity.
  bortezomib: Given IV
  lenalidomide: Given PO
Period: Overall Study
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Started | 53
Completed | 25
Not Completed | 28
Not completed — Adverse Event | 17
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Alternative therapy | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 67 [39 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Overall Response Defined as Complete Response and Partial Response
Description: Response is assessed by investigator according to International Working Group (IWG) criteria.
  A complete response requires disappearance of all evidence of disease. A partial response is a >/= 50% decrease in the sum of products of 6 largest dominant nodes or nodal masses as well as for splenic and hepatic nodules. No increase in size of nodes, liver or spleen and no new sites of disease.
Time Frame: Duration of treatment (assessed up to 6 years)
Measure: Number; unit: participants
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 53
participants | 21

2. Secondary Outcome: Incidence of Adverse Events
Description: Number of participants who experienced a maximum grade 3, 4 or 5 adverse event. The grading scales found in the revised NCI CTCAE version 4.0 was utilized for adverse event reporting
Time Frame: Duration of Treatment (up to 6 years)
Measure: Number; unit: participants
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 53
participants
  Grade 2 | 4
  Grade 3 | 29
  Grade 4 | 17
  Grade 5 | 1

3. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is defined as the time from study entry until progression or death due to any cause. The median TTP with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 53
years | 0.58 [0.29 to 1.15]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from study entry until death. The median OS with 95% CI was estimated using the Kaplan-Meier method..
Time Frame: Assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 53
years | 2.17 [1.15 to 4.58]

ADVERSE EVENTS:
Groups:
- Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy): lenalidomide: Given PO
Arm/Group | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 24/53
Other Adverse Events (participants affected / at risk) | 48/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy) (N=53)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 19 (23)
Mobitz type I (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Disease progression (General disorders) | 3 (3)
Edema limbs (General disorders) | 4 (4)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 15 (18)
Fever (General disorders) | 6 (7)
Abdominal infection (Infections and infestations) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Intraoperative complications (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (6)
Alkaline phosphatase increased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 3 (4)
Creatinine increased (Investigations) | 7 (8)
INR increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 11 (11)
Lymphocyte count decreased (Investigations) | 6 (8)
Neutrophil count decreased (Investigations) | 11 (12)
Platelet count decreased (Investigations) | 20 (24)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (6)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 8 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 11 (12)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (4)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (2)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (8)
Speech disorder (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (6)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antiangiogenesis Therapy, Enzyme Inhibitor Therapy) (N=53)
Hemoglobin decreased (Blood and lymphatic system disorders) | 38 (200)
Lymph node pain (Blood and lymphatic system disorders) | 2 (4)
Cardiac pain (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular trigeminy (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 2 (12)
Eye disorder (Eye disorders) | 2 (2)
Flashing vision (Eye disorders) | 1 (3)
Vision blurred (Eye disorders) | 5 (11)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (11)
Ascites (Gastrointestinal disorders) | 1 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 20 (76)
Diarrhea (Gastrointestinal disorders) | 22 (65)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 1 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (44)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (15)
Chills (General disorders) | 4 (7)
Edema limbs (General disorders) | 11 (19)
Fatigue (General disorders) | 37 (187)
Fever (General disorders) | 6 (7)
Flu-like symptoms (General disorders) | 1 (1)
General symptom (General disorders) | 1 (2)
Localized edema (General disorders) | 1 (2)
Pain (General disorders) | 2 (3)
Hypersensitivity (Immune system disorders) | 1 (2)
Immune system disorder (Immune system disorders) | 1 (35)
Bronchitis (Infections and infestations) | 3 (5)
Eye infection (Infections and infestations) | 2 (4)
Lip infection (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 4 (4)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (10)
Skin infection (Infections and infestations) | 4 (5)
Upper respiratory infection (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 11 (21)
Alkaline phosphatase increased (Investigations) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 11 (18)
Blood bilirubin increased (Investigations) | 3 (13)
Creatinine increased (Investigations) | 11 (17)
INR increased (Investigations) | 3 (5)
Laboratory test abnormal (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 18 (106)
Lymphocyte count decreased (Investigations) | 14 (49)
Neutrophil count decreased (Investigations) | 21 (156)
Platelet count decreased (Investigations) | 36 (203)
Weight loss (Investigations) | 8 (13)
Anorexia (Metabolism and nutrition disorders) | 16 (48)
Blood glucose increased (Metabolism and nutrition disorders) | 13 (67)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (16)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 10 (27)
Serum calcium decreased (Metabolism and nutrition disorders) | 9 (41)
Serum phosphate decreased (Metabolism and nutrition disorders) | 6 (28)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (12)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (9)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (7)
Ataxia (Nervous system disorders) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 14 (33)
Dysgeusia (Nervous system disorders) | 3 (6)
Extrapyramidal disorder (Nervous system disorders) | 2 (8)
Headache (Nervous system disorders) | 5 (9)
Neuralgia (Nervous system disorders) | 4 (13)
Neurological disorder NOS (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 7 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (281)
Sinus pain (Nervous system disorders) | 1 (2)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 5 (6)
Psychosis (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (3)
Testicular pain (Reproductive system and breast disorders) | 1 (6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (43)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (5)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (34)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 14 (27)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (5)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 6 (10)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 10 (16)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less